CLINICAL TRIAL: NCT06038604
Title: Psychosocial Support Program for Patients With Glioblastoma and Their Family Caregivers
Brief Title: Glioblastoma Psychosocial Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Glioblastoma Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110738
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial Support Intervention (Experimental): The psychosocial support intervention includes components such as logistical and practical support and self-care, strategies to manage cognitive changes, as well as strategies for effective communication when coping with glioblastoma.
  Interventions: Behavioral: Psychosocial Support Intervention

INTERVENTIONS:
Behavioral: Psychosocial Support Intervention — Participants will receive six weekly 60-minute sessions conducted by videoconference.

SUMMARY:
The goal of the study is to conduct a pilot test of the psychosocial support intervention with family caregivers and/or patients coping with glioblastoma.

DETAILED DESCRIPTION:
The specific aims of this study is to pilot test the psychosocial support program for patients with glioblastoma and/or their family caregivers. The investigators will recruit patient-caregiver dyads for the psychosocial support intervention; participants will have the choice whether to take part in the intervention as a dyad or individually given the variability of symptoms and progression of glioblastoma. The investigators will examine acceptability and feasibility of the intervention and examine whether participation in the program can help reduce distress and improve quality of life.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Patients who self-report a diagnosis of glioblastoma
* Age >18 years
* English Speaking

Exclusion Criteria:

* Lacks capacity for interview or is unable to provide informed consent
* Visual or hearing impairments or severe behavioral problems that preclude participation
* Too sick to participate

For caregivers:

Inclusion Criteria:

* Age >18 years
* English Speaking

Exclusion Criteria:

* Lacks capacity for interview or is unable to provide informed consent
* Visual or hearing impairments or severe behavioral problems that preclude participation
* Too sick to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete study participation | End of study (4-months)
  Completion of sessions by 70% of participants across a four-month period
Number of participants who complete post-intervention assessment | End of study (4-months)
  Completion of assessments by 70% of participants across a four-month period
Participants' satisfaction with treatment | End of study (4-months)
  Overall satisfaction rating for the psychosocial intervention with 70% of patients and caregivers reporting satisfaction. The Evaluation of Services measure will take the average of the item scores (0-4), with a mean of 3.0/4.0 as an indication of satisfaction

SECONDARY OUTCOMES:
Anxiety and depressive symptoms as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline; Post-intervention follow up (up to 4 months)
  The HADS will measure symptoms of anxiety and depression. The measure has 14 items (higher scores indicate higher distress).
General distress as measured by the Distress Thermometer | Baseline; Post-intervention follow up (up to 4 months)
  The Distress Thermometer will be used to measure general distress (higher scores indicate higher distress).
Functional well-being as measured by the Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline; Post-intervention follow up (up to 4 months)
  The functional well-being subscale of the FACT-G will be used to measure functional well-being (higher scores indicate higher functional well-being).
Caregiving efficacy as measured by the caregiver inventory | Baseline; Post-intervention follow up (up to 4 months)
  The caregiver inventory will be used to measure caregiving efficacy. The measure has 21 items (higher scores indicate higher levels of efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Laura S. Porter, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No